CLINICAL TRIAL: NCT02705482
Title: A Phase 1 Multicenter, Open-label, Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Antitumor Activity of MEDI0562 in Combination With Immune Therapeutic Agents in Adult Subjects With Advanced Solid Tumors
Brief Title: A Study to Evaluate MEDI0562 in Combination With Immune Therapeutic Agents in Adult Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6060C00002
Record Dates: First submitted 2015-09-22; First posted 2016-03-10 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Select Advanced Solid Tumors
Keywords: Advanced solid tumors; MEDI0562; durvalumab; tremelimumab; OX40; PD-L1; CTLA-4; immuno-oncology; Cancer
MeSH Terms: conditions — Diabetes Mellitus, Insulin-Dependent, 12; Neoplasms | interventions — tremelimumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: MEDI0562 and durvalumab (Experimental): MEDI0562 and durvalumab
  Interventions: Biological: MEDI0562; Biological: Durvalumab
- Arm B: MEDI0562 and tremelimumab (Experimental): MEDI0562 and tremelimumab
  Interventions: Biological: MEDI0562; Biological: Tremelimumab

INTERVENTIONS:
Biological: MEDI0562 — Subjects will remain on treatment until unacceptable toxicity, documentation of progressive disease (PD), or development of other reason for treatment discontinuation.
Biological: Tremelimumab — Subjects will remain on treatment until unacceptable toxicity, documentation of progressive disease (PD), or development of other reason for treatment discontinuation.
  Arms: Arm B: MEDI0562 and tremelimumab
Biological: Durvalumab — Subjects will remain on treatment until unacceptable toxicity, documentation of progressive disease (PD), or development of other reason for treatment discontinuation.
  Arms: Arm A: MEDI0562 and durvalumab

SUMMARY:
The purpose of this study is to evaluate MEDI0562 in combination with immune therapeutic agents in adult subjects with select advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1 multicenter, open-label study to evaluate the safety, pharmacokinetics, pharmacodynamics, immunogenicity, and antitumor activity of MEDI0562 in combination with immune therapeutic agents in adult subjects with select advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria:

1. Written and signed informed consent.
2. Age ≥ 18 years at the time of study entry.
3. Subjects must have received and have progressed, are refractory, or are intolerant to standard therapy appropriate for the specific tumor type. Subjects should not have received more than 3 prior lines of systemic therapy for recurrent or metastatic.
4. Subjects in the dose-escalation phase, must have histologic documentation of advanced solid tumors, excluding primary CNS tumors and hematologic malignancies.
5. Subjects in the dose-expansion phase, must have recurrent or metastatic disease solid tumors according to treatment arm as specified in the protocol.
6. Subjects who have received prior therapy with regimens containing CTLA 4, PD L1, or PD 1 antagonists are permitted to enroll if additional protocol criteria are met.
7. Subjects must have at least 1 lesion that is measurable using RECIST guidelines.
8. Subjects must consent to provide archived tumor specimens for correlative biomarker studies. In the setting where archival material is unavailable or unsuitable for use, subjects must consent and undergo fresh tumor biopsy.
9. All subjects are encouraged to consent to and provide both pretreatment and on treatment tumor biopsies.
10. ECOG Performance score of 0 or 1, unless protocol exceptions are met.
11. In the opinion of the investigator likely to complete ≥ 8 weeks of treatment.
12. Adequate hematologic, renal and hepatic function as determined by blood laboratory values.
13. At the time of Day 1 of the study, subjects with CNS metastases must have been treated and must be asymptomatic and meet the following:

    1. No concurrent treatment, inclusive of, but not limited to surgery, radiation, and/or corticosteroids
    2. At least 42 days without progression of CNS metastases as evidenced by magnetic resonance imaging (MRI) or computed tomography (CT) after last day of treatment
    3. At least 14 days since last dose of corticosteroids Note: Subjects with leptomeningeal disease or cord compression are excluded from the study.
14. Female subjects of childbearing potential who are sexually active with a non-sterilized male partner must use at least 1 highly effective method of contraception from screening, and must agree to continue using such precautions for 180 days after the final dose of investigational product.
15. Non-sterilized male subjects who are sexually active with a female partner of childbearing potential must use male condom plus, if locally available, spermicide from Day 1 and for 180 days after receipt of the final dose of investigational product.

Exclusion Criteria:

Any of the following would exclude the subject from participation in the study:

1. Prior treatment with TNFRSF agonists
2. Prior treatment with IMT for certain disease types may be restricted per protocol.
3. History of severe allergic reactions to any unknown allergens or any components of the study drug formulations
4. Active or prior documented autoimmune disease within the past 2 years.
5. Concurrent enrollment in another clinical study, unless it is an observational clinical study or the follow up period of an interventional study
6. Receipt of any conventional or investigational anticancer therapy not otherwise specified above within 28 days prior to the first dose
7. Any concurrent chemotherapy, IMT, or biologic or hormonal therapy for cancer treatment.
8. Unresolved toxicities from prior anticancer therapy.
9. Systemic therapeutic anticoagulation or daily aspirin dose exceeding 325 mg/per day.
10. Current or prior use of immunosuppressive medication within 14 days prior to the first dose of MEDI0562 with exceptions as per protocol.
11. History of primary immunodeficiency, solid organ transplantation, or tuberculosis
12. Test results indicating active infection with human immunodeficiency virus (HIV) or hepatitis B or C defined by positive serologic testing and confirmatory viral nucleic acid testing
13. Pregnant or breastfeeding women
14. Major surgery within 4 weeks prior to first dose of MEDI0562 or still recovering from prior surgery.
15. Other invasive malignancy within 2 years with the exception of protocol specified criteria
16. Any uncontrolled intercurent illness or condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Safety as defined by the presence of adverse events (AE), serious adverse events (SAE), and dose limiting toxicities (DLT). | From time of informed consent through 12 weeks after ending treatment with investigational product
  The primary endpoint is safety as assessed by presence of adverse event (AE), serious adverse event (SAE), and dose limiting toxicity (DLT).

SECONDARY OUTCOMES:
Preliminary Antitumor Activity:Best Overall Response | At approximately 3 time points through Day 113.
  The endpoints for assessment of antitumor activity include Best Overall Response (BOR) and will be based on all post-baseline disease assessments that occur prior to the initiation of subsequent anticancer therapy
Pharmacokinetics of MEDI0562/durvalumab or MEDI0562/tremelimumab: Cmax | To be assessed at approximately 12 clinic visits through Day 113
  The endpoints for assessment of PK of MEDI0562 and durvalumab or tremelimumab include individual MEDI0562, durvalumab, and tremelimumab concentrations at different time points after administration. PK parameters that may be modeled on these data include, but are not limited to, maximum observed concentration (Cmax).
Immunogenicity | At approximately 8 time points through Day 113.
  The endpoints for assessment of immunogenicity of MEDI0562, durvalumab, and tremelimumab include the number and percentage of subjects who develop detectable anti drug antibodies (ADAs).
Pharmacodynamic Activity | At approximately 12 time points through Day 113.
  The endpoints for assessment of pharmacodynamic activity include induction of proliferation markers in various lymphocyte populations and assessment of tumor-infiltrating lymphocytes (TILs) in tumor biopsy specimens.
Preliminary Antitumor Activity: Disease Control | At approximately 3 time points through Day 113.
  The endpoints for assessment of antitumor activity include disease control and is defined as CR, PR, or SD according to RECIST v1.1
Preliminary Antitumor Activity: Duration of Response | At approximately 3 time points through Day 113.
  The endpoints for assessment of antitumor activity include duration of response (DoR) and is defined as the duration from the first documentation of OR to the first documentation of disease progression or death due to any cause.
Preliminary Antitumor Activity: Progression-free Survival | At approximately 3 time points through Day 113.
  The endpoints for assessment of antitumor activity include progression-free survival (PFS) and is defined as the duration measured from the start of treatment with investigational product to the first documentation of disease progression or death due to any cause
Preliminary Antitumor Activity: Overall Survival | At approximately 3 time points through Day 113.
  The endpoints for assessment of antitumor activity include overall survival (OS) and is defined as the time from the start of treatment with Investigational Product until death due to any cause.
Pharmacokinetics of MEDI0562/durvalumab or MEDI0562/tremelimumab: AUC | To be assessed at approximately 12 clinic visits through Day 113
  The endpoints for assessment of PK of MEDI0562 and durvalumab or tremelimumab include individual MEDI0562, durvalumab, and tremelimumab concentrations at different time points after administration. PK parameters that may be modeled on these data include area under the concentration-time curve (AUC).
Pharmacokinetics of MEDI0562/durvalumab or MEDI0562/tremelimumab: Clearance | To be assessed at approximately 12 clinic visits through Day 113
  The endpoints for assessment of PK of MEDI0562 and durvalumab or tremelimumab include individual MEDI0562, durvalumab, and tremelimumab concentrations at different time points after administration. PK parameters that may be modeled on these data include clearance (CL).
Pharmacokinetics of MEDI0562/durvalumab or MEDI0562/tremelimumab: t½ | To be assessed at approximately 12 clinic visits through Day 113
  The endpoints for assessment of PK of MEDI0562 and durvalumab or tremelimumab include individual MEDI0562, durvalumab, and tremelimumab concentrations at different time points after administration. PK parameters that may be modeled on these data include terminal phase half-life (t½).
Preliminary Antitumor Activity: Objective Response | At approximately 3 time points through Day 113.
  The endpoints for assessment of antitumor activity include objective response (OR) and is defined as confirmed CR or confirmed PR based on RECIST v1.1
Preliminary Antitumor Activity: Time to Response | At approximately 3 time points through Day 113.
  The endpoints for assessment of Time to Response TTR and is defined as the time of first treatment to a subsequently confirmed CR or confirmed PR based on RECIST v1.1
Preliminary Antitumor Activity: Percent Change from Baseline | At approximately 3 time points through Day 113.
  The endpoints for assessment percent change from baseline in target lesion sum of diameters will be calculated at each adequate post baseline disease assessment with recorded measurement for all target lesions defined at baseline.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (9):
  - Research Site, Santa Monica, California
  - Research Site, Chicago, Illinois
  - Research Site, St Louis, Missouri
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, Huntersville, North Carolina
  - Research Site, Portland, Oregon
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
- Research Site, Villejuif, France
- Research Site, Amsterdam, Netherlands

REFERENCES:
- [Derived] Goldman JW, Piha-Paul SA, Curti B, Pedersen KS, Bauer TM, Groenland SL, Carvajal RD, Chhaya V, Kirby G, McGlinchey K, Hammond SA, Streicher K, Townsley DM, Chae YK, Voortman J, Marabelle A, Powderly J. Safety and Tolerability of MEDI0562, an OX40 Agonist mAb, in Combination with Durvalumab or Tremelimumab in Adult Patients with Advanced Solid Tumors. Clin Cancer Res. 2022 Sep 1;28(17):3709-3719. doi: 10.1158/1078-0432.CCR-21-3016. PMID 35699623